CLINICAL TRIAL: NCT01091402
Title: Autologous Serum Skin Test and Serum IL-18 Levels in Chronic Idiopathic Urticaria and Respiratory Allergic Diseases
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Other Study IDs: 1
Record Dates: First submitted 2010-03-23; First posted 2010-03-24 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2009-01

CONDITIONS: Urticaria; Respiratory Allergic Diseases
Keywords: autologous serum skin test, IL-18
MeSH Terms: conditions — Urticaria

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (4):
- chronic urticaria
  Interventions: Procedure: autologous serum skin test, serum IL-18
- asthma
  Interventions: Procedure: autologous serum skin test, serum IL-18
- seasonal allergic rhinitis
  Interventions: Procedure: autologous serum skin test, serum IL-18
- normal controls
  Interventions: Procedure: autologous serum skin test, serum IL-18

INTERVENTIONS:
Procedure: autologous serum skin test, serum IL-18

SUMMARY:
One of the proposed mechanisms in CU is autoimmunity. It was shown by a positive response to autologous serum skin test (ASST)in almost half of chronic urticaria (CU) patients. IL-18 also play a role in autoimmune disorders. The investigators aim was to investigate the relationship of ASST and IL-18 in CU and respiratory allergic diseases.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* chronic urticaria patients
* stable asthma patients
* allergic rhinitis patients with sensitized to pollens
* normal controls without atopic and skin disease.

Exclusion Criteria:

* unwillingness to the study
* other dermatological problems that could affect the skin test
* use of antihistamine drugs

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients from Outpatient clinic
Sampling Method: Non-Probability Sample
Dates: Start 2009-01

CONTACTS AND LOCATIONS:
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Turkey (Türkiye)